CLINICAL TRIAL: NCT00230009
Title: Brief Intervention in At-Risk First-time Mothers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Steven J. Ondersma, Associate Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NIDA-00516-3; K23DA000516 (NIH)
Record Dates: First submitted 2005-09-29; First posted 2005-09-30 (Estimated); Results first posted 2013-08-08 (Estimated); Last update posted 2013-08-08 (Estimated); Status verified 2013-08

CONDITIONS: Substance Use
Keywords: child abuse, child neglect, substance use, violence exposure, brief intervention
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Assessment only (No Intervention)
- Brief intervention session (Experimental)
  Interventions: Behavioral: Brief motivational intervention

INTERVENTIONS:
Behavioral: Brief motivational intervention
  Arms: Brief intervention session

SUMMARY:
Preliminary controlled trial of a brief intervention designed to reduce child maltreatment risk among low-income pregnant mothers. Foci will include major risk factors for maltreatment, including substance abuse, social isolation, depression, violence exposure, and maladaptive child-rearing attitudes/beliefs.

ELIGIBILITY:
Pregnant, expecting first child

Inclusion Criteria:

Receipt of public assistance (e.g., Medicaid, Food Stamps), ability to communicate in English

Exclusion Criteria:

Frank psychosis or other cognitive impairment

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2004-04; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Ondersma, Ph.D., Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

REFERENCES:
- [Background] Delaney-Black V, Covington C, Ondersma SJ, Nordstrom-Klee B, Templin T, Ager J, Janisse J, Sokol RJ. Violence exposure, trauma, and IQ and/or reading deficits among urban children. Arch Pediatr Adolesc Med. 2002 Mar;156(3):280-5. doi: 10.1001/archpedi.156.3.280. PMID 11876674
- [Background] Ondersma SJ, Chaffin MJ, Mullins SM, LeBreton JM. A brief form of the child abuse potential inventory: development and validation. J Clin Child Adolesc Psychol. 2005 Jun;34(2):301-11. doi: 10.1207/s15374424jccp3402_9. PMID 15901230
- [Background] Mullins SM, Bard DE, Ondersma SJ. Comprehensive services for mothers of drug-exposed infants: relations between program participation and subsequent child protective services reports. Child Maltreat. 2005 Feb;10(1):72-81. doi: 10.1177/1077559504272101. PMID 15611328
- [Background] Mullins SM, Suarez M, Ondersma SJ, Page MC. The impact of motivational interviewing on substance abuse treatment retention: a randomized control trial of women involved with child welfare. J Subst Abuse Treat. 2004 Jul;27(1):51-8. doi: 10.1016/j.jsat.2004.03.010. PMID 15223094

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants for this phase were recruited from a large prenatal care clinic affiliated with Wayne State University. Participants were either (a) approached while in the waiting area, or (b) identified via a participant database as being willing to be contacted regarding research studies.
Groups:
- Assessment Only: Brief assessment using Audio Computer Assisted Self Interview (A-CASI) technology to obtain the data only.
- Brief Intervention Session: Brief assessment using Audio Computer Assisted Self Interview (A-CASI) technology to obtain the data. Plus brief therapist-delivered motivational intervention, which was tied to the results of the A-CASI assessment (results from which were viewable immediately by the therapist).
Period: Single Session Intervention/Control
Arm/Group | Assessment Only | Brief Intervention Session
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0
Period: Follow-up
Arm/Group | Assessment Only | Brief Intervention Session
Started | 50 | 50
Completed | 19 | 24
Not Completed | 31 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Assessment Only | Brief Intervention Session | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 50 | 100
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 22.6 (4.4) | 23.6 (4.5) | 23.1 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 50 | 100
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Use
Description: Alcohol use was measured by looking at frequency of use in past 30 days with the Alcohol Use Disorders Identification Test (AUDIT), reported at the 3 month follow-up. The mean of each the control and intervention group was used. Frequency of use ranged from 0 to 5 for the follow-up sample. Higher scores mean more frequent use of the substance.
Time Frame: 3 month follow-up
Population: A total of 43 participants returned for follow-up and were the only participants analyzed on this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Assessment Only | Brief Intervention Session
Number analyzed (Participants) | 19 | 24
units on a scale | 1.37 (1.57) | 0.92 (1.35)

2. Primary Outcome: Drug Use
Description: Drug use was measured by looking at frequency of use in past 30 days with the Alcohol Use Disorders Identification Test (AUDIT), reported about marijuana use at the 3 month follow-up. The mean of each the assessment only and intervention group was used. Scores ranged from 0 to 13 for the follow-up sample. Higher scores mean more frequent use of the substance.
Time Frame: 3 month follow-up
Population: A total of 43 participants returned for follow-up and were the only participants analyzed on this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Assessment Only | Brief Intervention Session
Number analyzed (Participants) | 19 | 24
units on a scale | 1.89 (3.6) | 0.63 (1.76)

3. Primary Outcome: Child Abuse Potential
Description: Change score was calculated by taking the follow-up scores on the Brief Child Abuse Potential Inventory (BCAP) and subtracting the baseline score. The possible total score for the BCAP ranges from 0 to 24. Therefore, the possible range of scores for the change calculation (reported below) is -24 to +24. Higher scores indicate higher risk at the follow-up visit (worse outcome).
Time Frame: baseline and 3 month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Assessment Only | Brief Intervention Session
Number analyzed (Participants) | 19 | 24
units on a scale | -1.8 (5.8) | -2.4 (5.7)

4. Secondary Outcome: Depression
Description: Depression was measured by using the Center for Epidemiologic Studies Depression Scale (CES-D) at the 3 month follow-up. CES-D total scores can range from 0 to 60. Scores at 16 or higher indicate clinical significance. Higher scores represent higher risk for depression.
Time Frame: at 3 month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Assessment Only | Brief Intervention Session
Number analyzed (Participants) | 19 | 24
units on a scale | 19.74 (6.2) | 20.33 (6.5)

5. Primary Outcome: Treatment Engagement
Description: The number of participants who reported seeking outpatient substance abuse treatment since baseline (either at a treatment facility or through outpatient counseling).
Time Frame: at 3 month follow-up
Measure: Number; unit: participants
Arm/Group | Assessment Only | Brief Intervention Session
Number analyzed (Participants) | 19 | 24
participants | 0 | 1

ADVERSE EVENTS:
Arm/Group | Assessment Only | Brief Intervention Session
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

LIMITATIONS AND CAVEATS:
This study is limited by the relatively small sample size and the restriction to low-income, urban women, thus limiting generalizability to other populations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes